CLINICAL TRIAL: NCT06164015
Title: Association of Acquired Uterine Abnormalities With Recurrent Miscarriage
Brief Title: 3D Ultrasound to Assess in Recurrent Miscarriage
Acronym: 3D-ARM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2023/056
Record Dates: First submitted 2023-09-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Miscarriage
Keywords: Fibroids; Polyps; Adhesions; Adenomyosis; Endometrial blood flow
MeSH Terms: conditions — Abortion, Habitual; Leiomyoma; Polyps; Tissue Adhesions; Adenomyosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent Miscarriage group (study group): Group of women who have experienced 2 or more pregnancy loss of less than 24 weeks gestation.
  Interventions: Diagnostic Test: 3D Ultrasound scan with power Doppler angiography
- Fertile population group (control group): Group of women with proven fertility with at least one child born at full term
  Interventions: Diagnostic Test: 3D Ultrasound scan with power Doppler angiography

INTERVENTIONS:
Diagnostic Test: 3D Ultrasound scan with power Doppler angiography — The study group and the control group will be offered a 3D ultrasound scan as a part of this trial.

SUMMARY:
This observational study aims to compare the prevalence of acquired abnormalities of the uterus (fibroids, polyps, intrauterine adhesions, adenomyosis) in women who have recurrent miscarriages with the fertile population.

DETAILED DESCRIPTION:
High-quality studies including several meta-analyses have proven the association between congenital uterine anomalies and recurrent miscarriages. Nevertheless, there are limited studies evaluating the impact of acquired uterine anomalies on recurrent miscarriages.

This prospective observational study will aim to compare the prevalence of acquired uterine anomalies between the study group and the control group. The secondary aim will be to compare the Endometrial morphological features like endometrial volume, endometrial and sub-endometrial vascularity between the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Women between the age group of 18-40 years
2. Women who have had 2 or more pregnancy losses before 24 weeks of gestation - Study group.
3. Women who can provide documented informed consent
4. Women with proven fertility with at least one child - Control group

Exclusion Criteria:

1. Women with previous history of miscarriage/ extreme preterm delivery (before 28 weeks of gestation) will be excluded from the Control group.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender
Study Population: The professionals (clinicians, nurses) in the recurrent miscarriage clinic will identify the suitable study population. Suitable controls will be identified in the Gynae clinic,Gynae assessment unit,Gynaecology ward.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Acquired Uterine Anomalies | 24 months
  Primary outcome will be to compare the prevalence of acquired uterine anomalies (estimated as the proportion of anomalies diagnosed on 3D pelvic ultrasound) between study group and control group

SECONDARY OUTCOMES:
Endometrial thickness | 24 months
  measured by ultrasound (in mm)
Endometrial volume | 24 months
  measured by 3D ultrasound (in ml)
Endometrial blood flow indices (vascularisation index, flow index and vascularisation flow index) | 24 months
  All three indices as measured by 3D ultrasound using VOCAL software

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan YY, Jayaprakasan K, Tan A, Thornton JG, Coomarasamy A, Raine-Fenning NJ. Reproductive outcomes in women with congenital uterine anomalies: a systematic review. Ultrasound Obstet Gynecol. 2011 Oct;38(4):371-82. doi: 10.1002/uog.10056. PMID 21830244
- [Result] Carbonnel M, Pirtea P, de Ziegler D, Ayoubi JM. Uterine factors in recurrent pregnancy losses. Fertil Steril. 2021 Mar;115(3):538-545. doi: 10.1016/j.fertnstert.2020.12.003. PMID 33712099
- [Result] Dobson SJA, Jayaprakasan KM. Aetiology of recurrent miscarriage and the role of adjuvant treatment in its management: a retrospective cohort review. J Obstet Gynaecol. 2018 Oct;38(7):967-974. doi: 10.1080/01443615.2018.1424811. Epub 2018 Mar 20. PMID 29557233